CLINICAL TRIAL: NCT05938023
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled and Open Label Extension Study to Assess the Efficacy, Safety, and Pharmacokinetic Profile of of ATL1102 in Non-ambulatory Participants With Duchenne Muscular Dystrophy
Brief Title: A Study of ATL1102 or Placebo in Participants With Non-ambulatory Duchenne Muscular Dystrophy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study failed to meet its primary or secondary efficacy endpoints. In consultation with investigators, the sponsor determined that it is not in the best interests of patients for the study to continue.
Sponsor: Percheron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1102-DMD-Pre-CT03
Record Dates: First submitted 2023-06-05; First posted 2023-07-10 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Non-ambulatory; DMD
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo controlled treatment periods followed by open labelled treatment period
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ATL1102 25mg (Experimental): ATL1102 25mg administered subcutaneously once weekly
  Interventions: Drug: ATL1102 25mg
- ATL1102 50mg (Experimental): ATL1102 50mg administered subcutaneously once weekly
  Interventions: Drug: ATL1102 50mg
- Placebo (Placebo Comparator): Placebo is administered subcutaneously once weekly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATL1102 25mg — Dose and scheduled as specified in the Arm description
  Arms: ATL1102 25mg
Drug: ATL1102 50mg — Dose and scheduled as specified in the Arm description
  Arms: ATL1102 50mg
Drug: Placebo — Dose and scheduled as specified in the Arm description
  Arms: Placebo

SUMMARY:
This Phase IIb study is a two part, multicenter study to evaluate the efficacy, safety, pharmacokinetics and pharmacodynamics of ATL1102 in non-ambulant boys with Duchenne Muscular Dystrophy aged 10 to <18 years old. The study includes a randomised, double-blind, placebo-controlled treatment period (Part A), followed by an open labelled treatment period (Part B).

DETAILED DESCRIPTION:
This Phase IIb study is a two part, multicenter study to evaluate the efficacy, safety, pharmacokinetics and pharmacodynamics of ATL1102 and will enroll 45 non-ambulant boys with Duchenne Muscular Dystrophy (DMD) aged 10 to <18 years old.

During the 24 week randomised, double-blind, placebo-controlled treatment period (Part A) participants will be enrolled and randomised to receive either ATL1102 25mg, ATL1102 50mg or matched placebo in a 1:1:1 ratio given as a weekly subcutaneous injection.

Participants will then continue to the 24 week Open Labelled Treatment Period (Part B) and continue to receive ATL1102 25mg or ATL1102 50mg for a further 24 weeks. Participants on placebo in Part A will transition to ATL1102.

The study will consist of a 4 week screening period, 24 week randomised, double-blind, placebo-controlled treatment period (Part A), 24 week open label treatment period (Part B) and 16 week follow up period.

ELIGIBILITY:
Key Inclusion Criteria:

* Has a clinical diagnosis of DMD confirmed by validated genetic testing
* Is considered to be non-ambulatory, defined as unable to walk 10 meters without assistance or help at Screening.
* Male aged 10 to less than 18 years, at the time of Screening.
* Body weight of at least 25 kg at Screening.
* If receiving corticosteroid therapy, therapy was initiated at least six months prior to the baseline visit and a stable daily dose for at least 3 months prior to baseline
* Participant has a Performance of Upper Limb Module for DMD 2.0 (PUL 2.0) Entry Item A score ≥2.
* Able to perform spirometry and has sufficient Respiratory function defined as reproducible percent predicted FVC ≥50%.
* Has adequate cardiac function defined as left ventricular ejection fraction (LVEF) ≥45% by echocardiogram and if receiving cardiac medication, must be currently on a stable regimen and doses of cardiac therapy (at least 3 months prior to baseline Day 1)
* Participant and their parent/guardian/carer are willing and able to comply with scheduled visits, study medication administration and study procedures.

Key Exclusion Criteria:

* Participation in another clinical trial (non-interventional) or administration of any investigational product or experimental product within 12 weeks or 5 half-lives (whichever is longer) preceding Day 1.
* Exposure to more than 3 investigational products within the 12 months prior to Day 1.
* History of clinically significant bleeding or coagulation abnormalities or clinically significant abnormal coagulation parameters.
* Currently receiving antiplatelet or anticoagulant therapy or has taken medication with an antiplatelet or anticoagulant effect within 4 weeks prior Day 1
* Any evidence of clinically significant structural or functional heart abnormality (cardiomyopathy that is managed by ACEi or beta blockers is acceptable provided the LVEF inclusion criterion is met).
* Known history of or a positive test for hepatitis B surface antigen (HBsAg), hepatitis C (HCV) antibodies, human immunodeficiency virus (HIV) antibodies at Screening.
* Evidence of renal impairment and/or cystatin C >1.4 mg/L.
* Received a live vaccine (including intranasal influenza vaccine) within 4 weeks prior to Day 1 or planned live vaccination during the study period.
* Asthma (if requiring regular medication), bronchitis/chronic obstructive pulmonary disease (COPD), bronchiectasis, emphysema, pneumonia or the presence of any non-DMD respiratory illness that affects PEF and FVC or other respiratory measures.
* Requires day-time assisted mechanical or non-invasive ventilation (NIV) (night time NIV is permitted).
* Chronic use (daily intake >14 days), within one month of Day 1, of beta-2 agonists or any use of other bronchodilating medication (e.g., inhaled steroids, sympathomimetics, anticholinergics).
* Used carnitine, creatine, glutamine, oxatomide, idebenone or other forms of coenzyme Q10 or vitamin E or any other nutritional or antioxidant supplements or herbal medicines or anabolic steroids other than standard corticosteroids or puberty testosterone supplementation within 4 weeks of Day 1.
* Has an increased risk for opportunistic infections or systemic medical conditions resulting in significantly compromised immune system function

Ages: 10 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — DMD is a disease that predominantly affects males
Enrollment: 48 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Change in the Performance of Upper Limb (PUL) 2.0 score from baseline to Week 25 (blinded treatment period). | 25 weeks
  The PUL is an assessment used to evaluate the upper limb strength for individuals with DMD where a higher score indicates a better outcome with a minimum of 0 and a maximum score of 42
Change in the Performance of Upper Limb (PUL) 2.0 score from Week 25 to Week 49 (open label treatment period). | 49 weeks
  The PUL is an assessment used to evaluate the upper limb strength for individuals with DMD where a higher score indicates a better outcome with a minimum of 0 and a maximum score of 42
Change in the Performance of Upper Limb (PUL) 2.0 score from baseline to Week 49 (combined treatment period). | 49 weeks
  The PUL is an assessment used to evaluate the upper limb strength for individuals with DMD where a higher score indicates a better outcome with a minimum of 0 and a maximum score of 42
Safety measured by the incidence and frequency of adverse events, serious adverse events and suspected unexpected adverse events from baseline to Week 65 | 65 weeks
  An Adverse Event is any untoward medical occurrence in a participant and does not necessarily have to have a causal relationship with the intervention.

SECONDARY OUTCOMES:
Change in the grip strength of the hand from baseline to Week 25 using a handheld dynamometer tool (MyoGrip) (blinded treatment period). | 25 weeks
  The handheld dynamometer tool (MyoGrip) use strain gauge technology to measure the hand strength in Kilograms exerted by the participants with higher recordings indicating greater hand strength.
Change in the pinch strength of the fingers from baseline to Week 25 using handheld dynamometer tool (MyoPinch) (blinded treatment period). | 25 weeks
  The handheld dynamometer tool (MyoPinch) use strain gauge technology to measure the pinch strength of the fingers in Kilograms exerted by the participants with higher recordings indicating greater hand strength.
Change in the respiratory function assessed by Forced Vital Capacity (FVC) from baseline to Week 25 (blinded treatment period). | 25 weeks
  The percent predicted for Forced Vital Capacity (FVC%p) will be calculated at multiple timepoints after respiratory function is assessed using spirometry tests
Change in the respiratory function assessed by peak expiratory flow (PEF) from baseline to Week 25 (blinded treatment period). | 25 weeks
  The percent predicted for peak expiratory flow (PEF%p) will be calculated at multiple timepoints after respiratory function is assessed using spirometry tests
Change in the Paediatric Quality of Life (PedsQL™) questionnaire Duchenne Muscular Dystrophy (DMD) Module from baseline to Week 25 (blinded treatment period). | 25 weeks
  Health related quality of life is assessed by percentage of change in the score collected in the Paediatric Quality of Life (PedsQL™) Duchenne Muscular Dystrophy (DMD) Module for participants and parents at multiple timepoints. A higher score indicates a better health related quality of life with a minimum of 0 and a maximum score of 100.
Safety measured by the incidence and frequency of adverse events, serious adverse events and suspected unexpected adverse events from baseline to Week 25 (blinded treatment period). | 25 weeks
  An Adverse Event is any untoward medical occurrence in a participant and does not necessarily have to have a causal relationship with the intervention.
Maximum and minimum plasma concentration (Cmax and Cmin) for ATL1102 over multiple timepoints | 65 weeks
  Pharmacokinetic evaluation to evaluate dose response
Area under the plasma concentration time curve (AUC) for ATL1102 over multiple timepoints | 65 weeks
  Pharmacokinetic evaluation to evaluate dose concentration over time
Time to Cmax and Cmin for ATL1102 over multiple timepoints | 65 weeks
  Pharmacokinetic evaluation to evaluate concentration of ATL1102
The terminal half life for ATL1102 | 65 weeks
  Pharmacokinetic evaluation to evaluate the time for the ATL1102 concentration to reduce by half
Change in the grip strength of the hand from Week 25 to Week 49 using a handheld dynamometer tool (MyoGrip) (open label treatment period). | 49 weeks
  The handheld dynamometer tool (MyoGrip) use strain gauge technology to measure the hand strength in Kilograms exerted by the participants with higher recordings indicating greater hand strength.
Change in the pinch strength of the fingers from Week 25 to Week 49 using handheld dynamometer tool (MyoPinch) (open label treatment period). | 49 weeks
  The handheld dynamometer tool (MyoPinch) use strain gauge technology to measure the pinch strength of the fingers in Kilograms exerted by the participants with higher recordings indicating greater hand strength.
Change in the respiratory function assessed by Forced Vital Capacity (FVC) from Week 25 to Week 49 (open label treatment period). | 49 weeks
  The percent predicted for Forced Vital Capacity (FVC%p) will be calculated at multiple timepoints after respiratory function is assessed using spirometry tests
Change in the respiratory function assessed by peak expiratory flow (PEF) from Week 25 to Week 49 (open label treatment period). | 49 weeks
  The percent predicted for peak expiratory flow (PEF%p) will be calculated at multiple timepoints after respiratory function is assessed using spirometry tests
Change in the Paediatric Quality of Life (PedsQL) questionnaire Duchenne Muscular Dystrophy (DMD) Module from Week 25 to Week 49 (open label treatment period). | 49 weeks
  Health related quality of life is assessed by percentage of change in the score collected in the Paediatric Quality of Life (PedsQL™) Duchenne Muscular Dystrophy (DMD) Module for participants and parents at multiple timepoints. A higher score indicates a better health related quality of life with a minimum of 0 and a maximum score of 100.
Change in the grip strength of the hand from baseline to Week 49 using a handheld dynamometer tool (MyoGrip) (combined treatment period). | 49 weeks
  The handheld dynamometer tool (MyoGrip) use strain gauge technology to measure the hand strength in Kilograms exerted by the participants with higher recordings indicating greater hand strength.
Change in the pinch strength of the fingers from Baseline to Week 49 using handheld dynamometer tool (MyoPinch) (combined treatment period). | 49 weeks
  The handheld dynamometer tool (MyoPinch) use strain gauge technology to measure the pinch strength of the fingers in Kilograms exerted by the participants with higher recordings indicating greater hand strength.
Change in the respiratory function assessed by Forced Vital Capacity (FVC) from Baseline to Week 49 (combined treatment period). | 49 weeks
  The percent predicted for Forced Vital Capacity (FVC%p) will be calculated at multiple timepoints after respiratory function is assessed using spirometry tests
Change in the respiratory function assessed by peak expiratory flow (PEF) from baseline to Week 49 (combined treatment period). | 49 weeks
  The percent predicted for peak expiratory flow (PEF%p) will be calculated at multiple timepoints after respiratory function is assessed using spirometry tests
Change in the Paediatric Quality of Life (PedsQL) questionnaire Duchenne Muscular Dystrophy (DMD) Module from Baseline to Week 49 (combined treatment period). | 49 weeks
  Health related quality of life is assessed by percentage of change in the score collected in the Paediatric Quality of Life (PedsQL™) Duchenne Muscular Dystrophy (DMD) Module for participants and parents at multiple timepoints. A higher score indicates a better health related quality of life with a minimum of 0 and a maximum score of 100.

OTHER OUTCOMES:
Changes in lymphocyte populations to assess pharmacodynamic effects of ATL1102 from baseline to Week 57 | 57 weeks
  Lymphocyte population (cells/L) including cells expressing CD49d will be evaluated at multiple timepoints during the study utilizing chip cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Voit, Principal Investigator — UCL Great Ormond Street Institute of Child Health
Locations (13):
- Australia (3):
  - Royal Childrens Hospital, Melbourne
  - Queensland Children's Hospital, South Brisbane
  - The Children's Hospital at Westmead, Westmead
- UMHAT Aleksandrovska Neurology clinic, Sofia, Sofia, Bulgaria
- Serbia (2):
  - University Children's Hospital, Belgrade
  - Mother and Child Health Care Institute, Belgrade
- Turkey (Türkiye) (3):
  - Eskisehir Osmangazi Universitesi Tip Fakultesi, Eskişehir
  - Yeditepe University Hospital, Istanbul
  - Marmara University Pendik Training and Research Hospital, Pendik
- United Kingdom (4):
  - Birmingham Heartlands Hospital, Birmingham
  - The General Infirmary at Leeds, Leeds Teaching Hospital NHS Trust, Leeds
  - University College London (UCL) - Great Ormond Street Institute of Child Health (ICH), London
  - The Robert Jones and Agnes Hunt Orthopaedic Hospital, Oswestry

IPD SHARING:
Plan to Share IPD: No